CLINICAL TRIAL: NCT06339814
Title: Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol Applied to Caregivers of Children With Pediatric Brain Tumor: a Feasibility Study and a Pilot Randomized Group Treatment Trial.
Brief Title: Eye Movement Desensitization and Reprocessing Group Treatment for Caregivers of Pediatric Brain Tumor Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 05/23-CE
Record Dates: First submitted 2024-03-20; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Caregiver Burden
MeSH Terms: conditions — Caregiver Burden | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The study will be with two parallel branches, thus conforming to a Randomized Group Treatment Trial: Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol (those who will receive Eye Movement Desensitization and Reprocessing treatment plus the standard support) versus Treatment As Usual condition (those who will receive only standard support). The assessment will be performed at the moment of recruitment (T0), after the intervention for the Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol group and after 1 month for the Treatment As Usual condition (T1), and for both 2 months after T1 (T2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol (Experimental): Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol will receive Eye Movement Desensitization and Reprocessing treatment plus the standard support
  Interventions: Other: Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol; Other: Treatment As Usual
- Treatment As Usual group (Active Comparator): Treatment As Usual group will receive only standard support
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Other: Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol — An Eye Movement Desensitization and Reprocessing psychotherapist will hold the Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol sessions, dedicated to psychoeducation, imagery exercises, stabilization techniques and the reprocessing of traumatic events. The Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol will be composed of 4 sessions of 120 minutes each.
  Arms: Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol
Other: Treatment As Usual — Treatment As Usual condition will receive only standard support.

SUMMARY:
Caregivers of pediatric brain tumor survivors may develop high levels of psychological distress, mostly depression and anxiety, with effects comparable to those of a traumatic event. Several studies suggest that Eye Movement Desensitization and Reprocessing could be a promising treatment in similar clinical populations (i.e. adults with brain tumor), but it has never been used for caregivers of pediatric brain tumor. The aims of the present study will be to test the feasibility of the Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol for caregivers of pediatric brain tumor survivors in a clinical setting and to evaluate its effectiveness in decreasing the psychological distress in this population. The study will be monocentric, and with two parallel branches: the Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol group, who will receive a 4-session treatment, versus the Treatment as Usual condition, who will receive standard support. Emotional distress will be measured before the treatment, immediately after the end of it, and two months later (follow-up), by means of several clinical scales. Twenty-four subjects will be recruited for each group (caregivers and controls). Statistical analysis will be performed to test the effect of the intervention. If a positive outcome occurs, it could offer preliminary results about the validity of the Eye Movement Desensitization and Reprocessing in treating this population's difficulties.

DETAILED DESCRIPTION:
Pediatric cancer is a stressful life event, with a huge impact both on the diagnosed children and on their parents, comparable to that of a traumatic event. Caregivers of pediatric brain tumor survivors show several psychological difficulties, such as symptoms of anxiety, depression, and post-traumatic stress disorder. The presence of psychological distress throughout the oncological path of the child causes a long-term high burden impact, leading to an increased need for psychological support from the caregivers.

The Eye Movement Desensitization and Reprocessing has never been used for caregivers of pediatric brain tumor: neither individual nor Integrative Group Treatment Protocol. Hence, the aims of the present study are: (1) to test the feasibility of the Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol for caregivers of patients with pediatric brain tumor in a clinical setting; (2) to evaluate whether Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol is effective in decreasing psychological distress in caregivers.

Several studies suggest that Eye Movement Desensitization and Reprocessing could be a promising treatment for psychological distress, given the existing literature on caregivers of adult patients with brain tumor or dementia.

Design: The study will be monocentric, with two parallel branches, thus conforming to a Randomized Group Treatment Trial: Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol (those who will receive Eye Movement Desensitization and Reprocessing treatment plus the standard support) versus Treatment As Usual condition (those who will receive only standard support). The assessment will be performed at the moment of recruitment (T0), after the intervention for the Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol group and after 1 month for the Treatment As Usual condition (T1), and for both 2 months after T1 (T2).

Participants: Pediatric brain tumor caregivers and controls (24 subjects in each, 48 subjects in total) will be recruited at La Nostra Famiglia, IRCCS E. Medea, Bosisio Parini (LC), Italy. Inclusion criteria: being the primary caregivers of a patient with a diagnosis of brain tumor, with evidence of one or more traumatic events causing trauma related symptoms (Impact of Event Scale-Revised > 0, and Subjective Units of Distress > 5); being fluent in Italian and with at least three years of education. Exclusion criteria: Evidence of severe psychiatric disorders. Block randomization will be performed to ensure a balance in sample size across groups over time.

Caregivers' assessment will include: a data form to collect clinical and socio-demographic features (age, gender, educational level, occupation, type of pediatric brain tumor, treatments …), a feasibility questionnaire (only for the feasibility study), the Impact of Event Scale-Revised, the Subjective Units of Distress, the State-Trait Anxiety Inventory, the Beck Depression In-ventory, the Parenting Stress Index, the Caregiver Burden Inventory, and the Family Assessment Device 3.

Intervention: An Eye Movement Desensitization and Reprocessing psychotherapist will hold the Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol sessions, dedicated to psychoeducation, imagery exercises, stabilization techniques and the reprocessing of traumatic events. The Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol will be composed of 4 sessions of 120 minutes each. The number of the sessions has been chosen referring to the literature and based on the length of the hospitalization in the Institute. In the case of an emergency (e.g. increased number of Covid-19 cases), groups can also be held online. Supervision by an Eye Movement Desensitization and Reprocessing practitioner will be requested.

Analyses: (i) Spearman's correlations to test the relationship between clinical and socio-demographical variables; (ii) A series of generalized linear mixed models with clinical variables (outcomes of the psychological tests) as dependent variables, random intercept (grouped by subject) and with time (T0 versus T1 versus T2) and branch (Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol versus Treatment As usual) as fixed effect predictors to test the intervention.

If a decrease in the psychological symptoms occurs, it could offer preliminary results about the validity of the Eye Movement Desensitization and Reprocessing in alleviating the difficulties caregivers have in caring for pediatric BT survivor, easing the burden of an oncological disease with an unpredictable progression. Possible limitations of the study could include dropouts, the need for a wider sample for more rigorous results or a longer-term assessment (i.e. 6 months after the end of Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol ) to evaluate the stabilization of the positive effects.

ELIGIBILITY:
Inclusion Criteria:

* being the primary caregivers of a patient with a diagnosis of brain tumor,
* evidence of one or more traumatic events causing trauma related symptoms (Impact of Event Scale-Revised > 0, and Subjective Units of Distress > 5);
* being fluent in Italian
* with at least three years of education.

Exclusion Criteria:

* Evidence of severe psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Impact of Event Scale-Revised-Total score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Impact of Event Scale - Revised was designed as a measure of post-traumatic stress disorder symptoms, and is a short, easily administered self-report questionnaire. It can be used for repeated measurements over time to monitor progress and is best used for recent and specific traumatic events.
  Minimum-maximum value:0-88. Higher scores mean worse outcome.
Impact of Event Scale-Revised-Intrusion score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Impact of Event Scale - Revised was designed as a measure of post-traumatic stress disorder symptoms, and is a short, easily administered self-report questionnaire. It can be used for repeated measurements over time to monitor progress and is best used for recent and specific traumatic events.
  Minimum-maximum value:0-32;maximum mean score: 4. Higher scores mean worse outcome.
Impact of Event Scale-Revised-Avoidance score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Impact of Event Scale - Revised was designed as a measure of post-traumatic stress disorder symptoms, and is a short, easily administered self-report questionnaire. It can be used for repeated measurements over time to monitor progress and is best used for recent and specific traumatic events.
  Minimum-maximum value:0-32;maximum mean score: 4. Higher scores mean worse outcome.
Impact of Event Scale-Revised-Hyperarousal score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Impact of Event Scale - Revised was designed as a measure of post-traumatic stress disorder symptoms, and is a short, easily administered self-report questionnaire. It can be used for repeated measurements over time to monitor progress and is best used for recent and specific traumatic events.
  Minimum-maximum value:0-24;maximum mean score: 4. Higher scores mean worse outcome.
Subjective Units of Distress-Total Score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Subjective Units of Distress Scale is a tool for measuring the intensity of feelings and other internal experiences, such as anxiety, anger, agitation, stress or other painful feelings. The score ranges between 0 (no disturbance) and 10 (maximum perceived disturbance).
  Minimum-maximum value:0-10. Higher scores mean worse outcome.
State-Trait Anxiety Inventory-State anxiety score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The State-Trait Anxiety Inventory is a 40-item self-report scale that assesses separate dimensions of "state" and "trait" anxiety. Examples of what the the tool measures include feelings of apprehension, tension, nervousness, and worry.
  Minimum-maximum value: 20-80. Higher scores mean worse outcome.
State-Trait Anxiety Inventory-Trait anxiety score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The State-Trait Anxiety Inventory is a 40-item self-report scale that assesses separate dimensions of "state" and "trait" anxiety. Examples of what the the tool measures include feelings of apprehension, tension, nervousness, and worry.
  Minimum-maximum value: 20-80. Higher scores mean worse outcome.
Beck Depression Inventory-Total score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Beck Depression Inventory is a 21-item, multiple-choice inventory. Respondents are asked to rate each item based on four response choices according to the severity of the symptoms, ranging from the absence of a symptom to an intense level, during the past week.
  Minimum-maximum value: 0-63. Higher scores mean worse outcome.
Parenting Stress Index-Total score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Parenting Stress Index is used to measure the relative stress in the parent-child relationship. It can be used for parents of children up to 12 years.
  Minimum-maximum value: 36-180. Higher scores mean worse outcome.
Parenting Stress Index-Parental stress score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Parenting Stress Index is used to measure the relative stress in the parent-child relationship. It can be used for parents of children up to 12 years.
  Minimum-maximum value: 12-60. Higher scores mean worse outcome.
Parenting Stress Index-Dysfunctional interaction score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Parenting Stress Index is used to measure the relative stress in the parent-child relationship. It can be used for parents of children up to 12 years.
  Minimum-maximum value: 12-60. Higher scores mean worse outcome.
Parenting Stress Index-Hard child score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Parenting Stress Index is used to measure the relative stress in the parent-child relationship. It can be used for parents of children up to 12 years.
  Minimum-maximum value: 12-60. Higher scores mean worse outcome.
Stress Index for Parents of Adolescents-Total stress score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Stress Index for Parents of Adolescents is a screening and diagnostic instrument that identifies areas of stress in parent-adolescent interactions, allowing examination of the relationship of parenting stress to adolescent characteristics, parent characteristics, the quality of the adolescent-parent interactions, and stressful life circumstances. It can be used for parents of children between 11 and 19 years.
  Minimum-maximum value: 112-560. Higher scores mean worse outcome.
Stress Index for Parents of Adolescents-Life restrictions score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Stress Index for Parents of Adolescents is a screening and diagnostic instrument that identifies areas of stress in parent-adolescent interactions, allowing examination of the relationship of parenting stress to adolescent characteristics, parent characteristics, the quality of the adolescent-parent interactions, and stressful life circumstances. It can be used for parents of children between 11 and 19 years.
  Minimum-maximum value: 10-50. Higher scores mean worse outcome
Stress Index for Parents of Adolescents-Relationship with spouse/partner score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Stress Index for Parents of Adolescents is a screening and diagnostic instrument that identifies areas of stress in parent-adolescent interactions, allowing examination of the relationship of parenting stress to adolescent characteristics, parent characteristics, the quality of the adolescent-parent interactions, and stressful life circumstances. It can be used for parents of children between 11 and 19 years.
  Minimum-maximum value: 9-45. Higher scores mean worse outcome
Stress Index for Parents of Adolescents-Social alienation score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Stress Index for Parents of Adolescents is a screening and diagnostic instrument that identifies areas of stress in parent-adolescent interactions, allowing examination of the relationship of parenting stress to adolescent characteristics, parent characteristics, the quality of the adolescent-parent interactions, and stressful life circumstances. It can be used for parents of children between 11 and 19 years.
  Minimum-maximum value: 7-35. Higher scores mean worse outcome
Stress Index for Parents of Adolescents-Incompetence/guilt score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Stress Index for Parents of Adolescents is a screening and diagnostic instrument that identifies areas of stress in parent-adolescent interactions, allowing examination of the relationship of parenting stress to adolescent characteristics, parent characteristics, the quality of the adolescent-parent interactions, and stressful life circumstances. It can be used for parents of children between 11 and 19 years.
  Minimum-maximum value: 8-40. Higher scores mean worse outcome
Caregiver Burden Inventory-Time-dependence burden score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Caregiver Burden Inventory comprises 24 closed questions to assess the physical, psychological, emotional, social and financial problems experienced by family caregivers.
  Minimum-maximum value: 0-20. Higher scores mean worse outcome.
Caregiver Burden Inventory-Developmental burden score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Caregiver Burden Inventory comprises 24 closed questions to assess the physical, psychological, emotional, social and financial problems experienced by family caregivers.
  Minimum-maximum value: 0-20. Higher scores mean worse outcome.
Caregiver Burden Inventory-Physical burden score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Caregiver Burden Inventory comprises 24 closed questions to assess the physical, psychological, emotional, social and financial problems experienced by family caregivers.
  Minimum-maximum value: 0-16. Higher scores mean worse outcome.
Caregiver Burden Inventory-Social burden score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Caregiver Burden Inventory comprises 24 closed questions to assess the physical, psychological, emotional, social and financial problems experienced by family caregivers.
  Minimum-maximum value: 0-20. Higher scores mean worse outcome.
Caregiver Burden Inventory-Emotional burden score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The Caregiver Burden Inventory comprises 24 closed questions to assess the physical, psychological, emotional, social and financial problems experienced by family caregivers.
  Minimum-maximum value: 0-20. Higher scores mean worse outcome.
Family Assessment Device 3-Problem Solving score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The McMaster Family Assessment Device is a 60-item questionnaire that measures an individual's perceptions of his/her family.
  Minimum-maximum value: 6-24. Higher scores mean worse outcome.
Family Assessment Device 3-Communication score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The McMaster Family Assessment Device is a 60-item questionnaire that measures an individual's perceptions of his/her family.
  Minimum-maximum value: 6-40. Higher scores mean worse outcome.
Family Assessment Device 3-Roles score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The McMaster Family Assessment Device is a 60-item questionnaire that measures an individual's perceptions of his/her family.
  Minimum-maximum value: 6-44. Higher scores mean worse outcome.
Family Assessment Device 3-Affective Responsiveness score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The McMaster Family Assessment Device is a 60-item questionnaire that measures an individual's perceptions of his/her family.
  Minimum-maximum value: 6-24. Higher scores mean worse outcome.
Family Assessment Device 3-Affective Involvement score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The McMaster Family Assessment Device is a 60-item questionnaire that measures an individual's perceptions of his/her family.
  Minimum-maximum value: 6-28. Higher scores mean worse outcome.
Family Assessment Device 3-Behavior Control score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The McMaster Family Assessment Device is a 60-item questionnaire that measures an individual's perceptions of his/her family.
  Minimum-maximum value: 6-36. Higher scores mean worse outcome.
Family Assessment Device 3-General Functioning score | at the moment of recruitment (T0), after 1 month (T1), and 2 months after T1 (T2) for both groups
  The McMaster Family Assessment Device is a 60-item questionnaire that measures an individual's perceptions of his/her family.
  Minimum-maximum value: 6-48. Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Chiara Oprandi, Principal Investigator — IRCCS Eugenio Medea
Locations (1):
- IRCCSEMedea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No